CLINICAL TRIAL: NCT03074214
Title: Study of Prognostic Value of Copeptin for Myocardial Infarct Size and 6-month Prognosis in Patients With ST-elevation Myocardial Infarction Undergoing Percutaneous Coronary Intervention: GOOD I Study
Brief Title: Prognostic Value of Copeptin for Infarct Size and Prognosis in Patients With ST-elevation Myocardial Infarction
Acronym: GOODI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, YU Tong-tong, Principal Investigator, Shengjing Hospital
Other Study IDs: 2016PS373K
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: copeptin; myocardial infarct size; prognosis; ST-elevation myocardial infarction; percutaneous coronary intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Diabetes Insipidus | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A venous blood sample will be collected at before, immediately after, and 3 days after PPCI and 6-month visit for biomarker analysis and storage for future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI patients receiving PCI: patients with STEMI receiving percutaneous coronary intervention
  Interventions: Procedure: percutaneous coronary intervention

INTERVENTIONS:
Procedure: percutaneous coronary intervention — All STEMI patients enrolled will at first receive "Device"(such as: stent or balloon) treatment for their coronary artery.

SUMMARY:
ST-elevation myocardial infarction (STEMI) has a serious health threaten to population. PCI, which can timely restore the blood flow to the ischemic myocardium, is a well-proved measure in STEMI management. However, the process of the restoration can induce injury. The phenomenon is defined as ischemia/reperfusion (I/R) injury. The studies indicate that I/R injury accounts for up to 50% of the final myocardial infarct size. However, previous attempts to target known mediators of myocardial I/R injury in patients have been disappointing, leading to calls for a reevaluation of factors affecting myocardial I/R injury [1]. Arginine vasopressin (AVP), that response to acute illness, is unstable and cleared rapidly from the circulation. However, copeptin, the C-terminal portion of provasopressin, is released in equimolar amounts to AVP and is easy to determine. So, copeptin can be a surrogate marker for AVP secretion. Recently, copeptin was found to serve as a potential prognostic biomarker in heart failure and acute myocardial infarction (AMI). AMI can activate the AVP axis, which have a causative role in the evolution of heart failure. Increasing copeptin was shown to correlate with myocardial remodeling, mortality and morbidity. In patients with STEMI, myocardial infarct size is a stronger outcome predictor than LV function, and is related to LV remodeling, which often indicates a significant worse prognosis after AMI. As the gold standard for characterisation of cardiac structure and function, cardiac magnetic resonance (CMR) parameters can serve as surrogate end points in clinical trials of STEMI. We hypothesised that plasma copeptin values, tested before and after PCI, are related to myocardial infarct size, myocardial function both and outcomes at baseline and 6 months follow-up as assessed by CMR in patients with STEMI.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is a major concern in public health in China. Ischemia/reperfusion injury cripples the treatment effect of reperfusion management, and increases the final myocardial infarct size. Copeptin is related to the prognosis of heart failure and AMI, and may be a potential prognostic biomarker for myocardial infarct size, myocardial function and outcomes in patients with STEMI undergoing PCI.This study will enroll consecutive STEMI patients undergoing PCI, who meet the inclusion and exclusion criteria, in a large-scale hospital in Northeast China. After obtaining an informed consent, blood samples will be drawn at the time of before, immediately after, and 3 days after PPCI. They will be collected in EDTA tubes and centrifuged for 10 min at 2000 g within 0.5 h. Plasma will be stored at -80°C until analysis. Plasma copeptin concentrations will be determined by a commercially available automated immunofluorescent assay (R&D Systems Inc. Minneapolis, USA). And other information about symptoms, functioning, quality of life, medical care, demographic characteristics, medical history, clinical features, diagnostic tests, medications and procedural data will be also collected. Baseline CMR will be performed 3-5 days after PPCI. All scans were performed on a 3.0 Tesla scanner. At 1 month, 3 month, and 12 month after discharge, participants will receive a follow-up by phone. At 6 month after discharge, participants will return to the clinic for follow up visits, and a face-to-face interview will be conducted to get information about clinical events, symptoms, functioning, quality of life, and medical care during the recovery period. Follow-up CMR scan will be conducted. Follow-up blood samples will be drawn for testing copeptin.

Sample Size Calculation A study size analysis was performed using PASS (version 11.0.4, 2011, NCSS, LLC, USA). In a previous study, the 90-day primary composite end point of all-causes death, ventricular fibrillation, cardiogenic shock, and congestive heart failure requiring rehospitalization or an emergency room visit through 90 days was 10.3% in STEMI patients undergoing PCI. [1] Although available data for detecting clinically relevance between copeptin and prognosis in STEMI patients undergoing PCI was limited, a previous study demonstrated that a high concentration (quartile 4 vs. quartiles 1 to 3) of copeptin identified an increased risk of CV death or HF (HR:2.80,95%CI:2.24-3.51,P<0.001). [2] When the ratio between groups1 and 2 is 3:1, an overall sample size of 275 subjects, of which 207 are in group 1 and 68 are in group 2, achieves 90% power at a 0.0500 significance level to detect a difference of 0.1280 between 0.9290 and 0.8010--the proportions surviving in groups 1 and 2, respectively. The proportion of patients lost during follow up was 0.1000.

ELIGIBILITY:
Inclusion Criteria:

1. chest pain present less than 12 hours from onset of pain to time of catheterization;
2. significant ST-segment elevation (at least 0.1 mV in two or more standard leads or at least 0.2 mV in two or more contiguous precordial leads) or a new left bundle branch block;
3. receiving primary PCI.

Exclusion Criteria:

1. Patients with conditions other than STEMI that could cause increased copeptin levels, such as renal dysfunction (eGFR<30 ml/min), liver failure, respiratory tract infection, stroke, sepsis, hyponatremia (Serum sodium concentration<135mmol/L), central diabetes insipidus or malignancy;
2. Patients with contraindications to perform cardiac magnetic resonance;
3. Patients with cardiogenic shock (Killip class IV);
4. Patients in whom reperfusion therapy failed;
5. Patients who were referred for emergency coronary artery bypass grafting (CABG) in view of unfavourable coronary anatomy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 275 patients with STEMI receiving PPCI in department of Cardiology, Shengjing Hospital of China Medical University from March 1, 2017 to February 28, 2019
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 6 months
  Composite of MACE including cardiac death, non-fatal myocardial reinfarction, unplanned repeat revascularization, congestive heart failure or angina requiring rehospitalization or an emergency room visit, ventricular fibrillation or ventricular tachycardia with hemodynamic instability

SECONDARY OUTCOMES:
All-cause death | 6 months
  All-cause death
Cardiac death | 6 months
  Cardiac death
unplanned repeat revascularization | 6 months
  unplanned repeat revascularization which included any unplanned repeat PCI or surgical bypass of target or non-target vessels
congestive heart failure requiring rehospitalization or an emergency room visit | 6 months
  congestive heart failure requiring rehospitalization or an emergency room visit
angina requiring rehospitalization or an emergency room visit | 6 months
  angina requiring rehospitalization or an emergency room visit
ventricular fibrillation or severe ventricular tachycardia | 6 months
  ventricular fibrillation or severe ventricular tachycardia with hemodynamic instability occurring more than 2 hours after PCI
acute heart failure during the index hospitalization | 6 months
  acute heart failure during the index hospitalization
in-stent stent thrombosis | 6 months
  acute, subacute or chronic in-stent stent thrombosis
contrast-induced nephropathy | 6 months
  Contrast-induced nephropathy was deﬁned as an increase in serum creatinine concentration ≥0.5 mg/dl (44.2 mmol/l) or ≥25% above baseline 72 h after exposure to the contrast medium.
ischemia stroke | 6 months
  ischemia stroke was defined as an acute event of non-hemorrhagic cerebrovascular origin causing focal or global neurologic dysfunction lasting >24 h, which was confirmed by both clinical and radiographic criteria.
Bleeding Academic Research Consortium Definition for Bleeding: type 3 or 5 | 6 months
  Bleeding Academic Research Consortium Definition for Bleeding: Type 3 Type 3a Overt bleeding plus hemoglobin drop of 3 to 5 g/dL* (provided hemoglobin drop is related to bleed) Any transfusion with overt bleeding Type 3b Overt bleeding plus hemoglobin drop 5 g/dL* (provided hemoglobin drop is related to bleed) Cardiac tamponade Bleeding requiring surgical intervention for control (excluding dental/nasal/skin/hemorrhoid) Bleeding requiring intravenous vasoactive agents;Type 3c Intracranial hemorrhage (does not include microbleeds or hemorrhagic transformation, does include intraspinal) Subcategories confirmed by autopsy or imaging or lumbar puncture Intraocular bleed compromising vision Type 5: fatal bleeding Type 5a Probable fatal bleeding; no autopsy or imaging confirmation but clinically suspicious Type 5b Definite fatal bleeding; overt bleeding or autopsy or imaging confirmation
Seattle angina questionnaire (SAQ) | 6 months
  Seattle angina questionnaire (SAQ)
Quality of life (EQ-5D) | 6 months
  Quality of life (EQ-5D)
Depression (PHQ-8) | 6 months
  Depression (PHQ-8)
Stress (Chinese 14-item PSS) | 6 months
  Stress (Chinese 14-item PSS)
Cognitive function (MMSE) | 6 months
  Cognitive function (MMSE)
myocardial infarct size | 6 months
  myocardial infarct size

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoqing Su, Doctor, Study Chair — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No
We will not share IPD to protect our data very well.

REFERENCES:
- [Background] Ellis SG, Tendera M, de Belder MA, van Boven AJ, Widimsky P, Janssens L, Andersen HR, Betriu A, Savonitto S, Adamus J, Peruga JZ, Kosmider M, Katz O, Neunteufl T, Jorgova J, Dorobantu M, Grinfeld L, Armstrong P, Brodie BR, Herrmann HC, Montalescot G, Neumann FJ, Effron MB, Barnathan ES, Topol EJ; FINESSE Investigators. Facilitated PCI in patients with ST-elevation myocardial infarction. N Engl J Med. 2008 May 22;358(21):2205-17. doi: 10.1056/NEJMoa0706816. PMID 18499565
- [Background] O'Malley RG, Bonaca MP, Scirica BM, Murphy SA, Jarolim P, Sabatine MS, Braunwald E, Morrow DA. Prognostic performance of multiple biomarkers in patients with non-ST-segment elevation acute coronary syndrome: analysis from the MERLIN-TIMI 36 trial (Metabolic Efficiency With Ranolazine for Less Ischemia in Non-ST-Elevation Acute Coronary Syndromes-Thrombolysis In Myocardial Infarction 36). J Am Coll Cardiol. 2014 Apr 29;63(16):1644-53. doi: 10.1016/j.jacc.2013.12.034. Epub 2014 Feb 13. PMID 24530676